CLINICAL TRIAL: NCT04651166
Title: Effect of Prophylactic Tranexamic Acid on Bleeding Outcomes for Dilation and Evacuation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Hawaii (Other)
Collaborators: Society of Family Planning (Other)
Responsible Party: Principal Investigator, Marit Pearlman Shapiro, Complex Family Planning Fellow, University of Hawaii
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RA-2020-050
Record Dates: First submitted 2020-11-25; First posted 2020-12-03 (Actual); Last update posted 2023-09-06 (Actual); Status verified 2023-08

CONDITIONS: Abortion; Dilation and Evacuation; Hemorrhage; Blood Loss
MeSH Terms: conditions — Dilatation, Pathologic; Hemorrhage | interventions — Tranexamic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo (Placebo Comparator): 100mL saline or lactated ringer without tranexamic acid added given intravenously over 10 minutes at start of procedure
  Interventions: Drug: Placebo
- Active Comparator (Active Comparator): 1g tranexamic acid mixed in 100mL saline or lactated ringer given intravenously over 10 minutes at start of procedure
  Interventions: Drug: Tranexamic acid

INTERVENTIONS:
Drug: Tranexamic acid — 1g tranexamic acid mixed in 100mL saline or lactated ringer
  Arms: Active Comparator
Drug: Placebo — 100mL saline or lactated ringers
  Arms: Placebo

SUMMARY:
Prophylactic tranexamic acid has shown been shown to reduce maternal mortality from postpartum hemorrhage with no adverse effects, but has not been studied to reduce bleeding complications with dilation and evacuation (D&E). We propose a randomized, double-blinded, placebo-controlled pilot study to determine whether routine use of intravenous (IV) tranexamic acid will decrease the need for interventions to control bleeding at the time of D&E at 16 to 24 weeks gestation.

ELIGIBILITY:
Inclusion Criteria:

* Requesting pregnancy termination
* Intrauterine pregnancy at 16 to 24 weeks gestation
* Participants must be willing and capable of giving informed consent and able to understand and sign written consents in English.

Exclusion Criteria:

* History of thromboembolic events (i.e. deep vein thrombosis, stroke, pulmonary embolism)

Min Age: 14 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2022-02-15 (Actual); Primary Completion 2023-07-27 (Actual); Study Completion 2023-07-27 (Actual)

PRIMARY OUTCOMES:
Intervention to control blood loss | At time of procedure
  Rate at which providers perform interventions to control blood loss during D&E procedures

CONTACTS AND LOCATIONS:
Overall Officials: Marit Pearlman Shapiro, Principal Investigator — University of Hawaii
Locations (1):
- Queens Medical Center, Honolulu, Hawaii, United States

IPD SHARING:
Plan to Share IPD: No